CLINICAL TRIAL: NCT01549145
Title: Sub-chronic Neurostimulation Delivered in the Middle Ear for Tinnitus Suppression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EstimME Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EST-01-IL; NCT01139554 (obsolete NCT alias)
Record Dates: First submitted 2012-03-06; First posted 2012-03-09 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Tinnitus
Keywords: Severe; Ongoing; Unilateral; present for more than 6 months
MeSH Terms: conditions — Tinnitus; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NIMBUS multifunctional stimulator (Experimental): A Multifunctional Stimulator (Nimbus by Newmedic, Hemodia) for clinical use. The stimulator is also dedicated for Electrical Promontory Stimulation (EPS)
  Interventions: Device: Nimbus Multifunctional Stimulator

INTERVENTIONS:
Device: Nimbus Multifunctional Stimulator — A Multifunctional Stimulator (Nimbus by Newmedic, Hemodia) for clinical use. The stimulator is also dedicated for Electrical Promontory Stimulation (EPS)

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of applying electrical stimulation on the promontorium (EPS) for the suppression of tinnitus in a sub-chronic stimulation regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Total score on the Handicap Inventory (THI) of at least 40.
2. Visual scale over 5.
3. Tinnitus origin is peripheral (related to long term noise exposure, or to a sudden exposure to a very loud noise etc.)
4. Tinnitus is on-going; present for more than 50% of the time over the past 12 months.
5. Unilateral tinnitus
6. Tinnitus prevalent at least 12 months.
7. Willingness to abstain from part taking in other, non-study procedures indicated to lessen tinnitus and/or its perception.
8. Willing and able to refrain from engaging in activities or work involving loud noise exposure.
9. Male or females 18-60 years of age

Exclusion Criteria:

1. Prior history of sudden hearing loss and/or fluctuating hearing levels.
2. Tinnitus prevalent more than 3 years.
3. History of frequent middle ear infections
4. Patient under immunosuppressant therapy
5. Auditory nerve damage.
6. Vestibular Schwannoma
7. Cochlear implant.
8. Pregnant or lactating.
9. Developmental disability or cognitive impairment that would make it difficult for the subject to partake in the clinical study, including adequate comprehension of the informed consent form and ability to record the necessary measurements.
10. Involvement in litigation and/or a worker's compensation claim and/or receiving disability benefits related to tinnitus and/or hearing loss.
11. Not being physically or geographically capable of returning for scheduled follow-up visits.
12. Any physical, psychological, or emotional disorder that would interfere with the planned surgical operations
13. Mentally retarded, developmentally delayed or suffering from organic brain dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Efficacy | 2 months
  Study efficacy evaluations will be based on the analysis of pre and post procedure tinnitus severity characteristics (THI, MML, Pitch matching and VAS values).

SECONDARY OUTCOMES:
Safety | 2 months
  Safety evaluations will be based on the observation for the reporting of any adverse events occurring during the study and up to the 30 days follow-up visit Occurrence of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel